CLINICAL TRIAL: NCT01900951
Title: Phase 2 Study of Temozolomide as Maintenance Therapy After Initial Induction Chemotherapy in Small Cell Lung Cancer
Brief Title: Temozolomide as Maintenance Therapy in Small Cell Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, yihu, chief physician, Chinese PLA General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TMS-01
Record Dates: First submitted 2013-07-11; First posted 2013-07-17 (Estimated); Last update posted 2016-01-26 (Estimated); Status verified 2016-01

CONDITIONS: Carcinoma, Small Cell
Keywords: Small cell lung cancer; temozolomide; Maintenance chemotherapy
MeSH Terms: conditions — Carcinoma, Small Cell; Small Cell Lung Carcinoma | interventions — Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Temozolomide (Experimental): Patients in the study will receive the following for the duration of the study:First-line chemotherapy according to the NCCN guidelines. The study will consist of 21-day cycles, to a maximum of 6 cycles of therapy for the first-line chemotherapy. After first-line treatment, temozolomide will be given alone as maintenance therapy in all patients who have achieved study entry hematologic criteria and who do not have progressive disease or severe toxicity. During temozolomide maintenance therapy, patients will receive temozolomide at 150mg/m2/d for 5 days of a 28-day cycle orally daily. Temozolomide maintenance therapy will continue until progressive disease or irreversible toxicity occurs.
  Re-staging will be performed every 2 cycles (every 8 weeks) during the study
  Interventions: Drug: Temozolomide

INTERVENTIONS:
Drug: Temozolomide

SUMMARY:
Temozolomide, a nonclassic oral alkylating agent, may delay progression in sequence with chemotherapy. This phase II trial was designed to evaluate the role of Temozolomide following 4 or 6 cycles of first-line treatment in patients with newly diagnosed SCLC.

DETAILED DESCRIPTION:
Subjects will receive standard of care treatment for SCLC with added treatment of maintenance temozolomide. Efficacy and safety of temozolomide and one year survival and time to progression of patients will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Cytologically and/or histologically confirmed small-cell lung cancer with extensive-stage disease
* Patients must have measurable disease, this can include brain metastases
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-1
* Adequate bone marrow function, as defined by: absolute neutrophil count (ANC) >1,500/µL; platelets >100,000/µL; hemoglobin >=9.0 g/dL
* Normal organ function, defined as follows: aspartate aminotransferase (AST) and alanine aminotransferase (ALT) <=2.5 × the upper limit of normal (ULN), or AST and ALT <=5 × the ULN if liver function abnormalities are due to underlying malignancy; total serum bilirubin <=1.5 × the ULN; serum creatinine <=1.5 × the ULN
* Women of childbearing potential and men with partners of childbearing potential must agree to use a form of birth control that is acceptable to their physician to prevent pregnancy during treatment
* Patients must be informed of the investigational nature of this study and sign an informed consent form

Exclusion Criteria:

* Patients who are pregnant or breastfeeding
* Patients receiving other investigational agents
* Patients with leptomeningeal involvement
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, or psychiatric illness/social situations that would limit compliance with study requirements
* Acquired Immune Deficiency Syndrome (AIDS) based upon current CDC definition or HIV-positive patients on combination antiretroviral therapy. However, HIV testing is not required for entry into this protocol. The need to exclude patients with AIDS from this protocol is necessary because these patients are at increased risk of lethal infections when treated with marrow- suppressive therapy. Excluding patients on HAART is necessary due to the potential for pharmacokinetic interactions with temozolomide.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2013-01; Primary Completion 2016-02 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
One-year progress free survival | 18 months
  The Percentage of Patients Who Are Progress Free One Year After Completing Protocol Treatment

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | 18 months
  the Percentage of Patients Who Experience an Objective Benefit From Treatment
Safety | 18 months
  Number of Participants with Adverse Events as a Measure of Safety and Tolerability
time to progression | from the start date of treatment until the date of occurrence of progressive disease
  the interval between the start date of treatment and the date of occurrence of progressive disease

CONTACTS AND LOCATIONS:
Overall Officials: yi hu, M.D., Study Chair — Chinese PLA General Hospital
Locations (1):
- PLA general hospital, Beijing, Beijing Municipality, China